CLINICAL TRIAL: NCT02317601
Title: Preoperative Single-high Dose Glucocorticoid for Patients Undergoing Hip Fracture Surgery and the Effect on Postoperative Delirium.
Brief Title: Preoperative Single Glucocorticoid Hip Fracture Hip Fracture Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Christopher Clemmesen, MD, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2014-002492-29; 2014-002492-29 (EudraCT Number)
Record Dates: First submitted 2014-11-27; First posted 2014-12-16 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-07

CONDITIONS: Delirium - Postoperative; Stress, Physiological
MeSH Terms: conditions — Emergence Delirium | interventions — Methylprednisolone Hemisuccinate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methylprednisolone sodium succinate (Active Comparator): 125 mg iv, as single dose, preoperative.
  Interventions: Drug: methylprednisolone sodium succinate
- physiological saline (Placebo Comparator): 5 mL of Sodium-Chloride 9 mg/ml, Fresenius Kabi
  Interventions: Drug: placebo saline

INTERVENTIONS:
Drug: methylprednisolone sodium succinate — Single dose Intravenous
  Other Names: Solu-medrol Product Code 52245
  Arms: Methylprednisolone sodium succinate
Drug: placebo saline
  Arms: physiological saline

SUMMARY:
The Study is a double-blinded, randomized, placebo-controlled trials. The Objective is to investigate the effect of single-high-dose glucocorticoid on surgical stress response and postoperative delirium among Elderly hip Fracture Patients undergoing surgery.

DETAILED DESCRIPTION:
Patients with Hip Fracture are exposed for two traumas that can trigger a stress response. The first is the fall that causes the Fracture. The second is the surgery. In this study the intervention is dispensed early in the disease course - as soon as the Fracture has been diagnosed and booked for surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgery for hip fracture
* Informed signed consent
* Danish speaking

Exclusion Criteria:

* Allergies towards contents of Solu-Medrol
* Insulin dependent diabetes
* Glaucoma
* In treatment for cancer disease
* Positive HIV, Hepatitis b or C status
* Lack of informed consent (eq. Severe dementia, coma, and others)
* Current treatment with systemic glucocorticoids (pr.os or intravenous) Immunoinflammatory disease (Except topical treated skin disease and respiratory disease)
* Current Immunosuppressive treatment
* Unable to participate in CAM-S measurement
* Peptic ulcera

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 122 (Actual)
Dates: Start 2014-12; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Post operative delirium measured with Confusion Assessment Method severity measure CAM-S | 3 first post operative days
  Post operative delirium measured with Confusion Assessment Method severity measure CAM-S

SECONDARY OUTCOMES:
Post operative delirium incidents measured by CAM-S | 3 days
  Incidents of delirium measured by CAM-S
Patient mobility measured by Cumulated Ambulation Score (CAS) | 3 first operative days
  Physiotherapy
The degree of inflammatory response measured by biomarker in the blood (suPAR, Interleukin 6, and others) | 4 days
  Biomarker
Post operative Fatigue measured with a patient fatigue self-assessment 0-4. (Verbal rating scale) 0=no fatigue, 1=mild, 2 = moderate, 3 = severe, 4 = excruciating (in bed because of fatigue). | 3 first postoperative days
  Measured with a patient fatigue self-assessment 0-4. (Verbal rating scale) 0=no fatigue, 1=mild, 2 = moderate, 3 = severe, 4 = excruciating (in bed because of fatigue).
Psychiatric medications (total amount/use of psychiatric medications) | 3 post-OR days
  The total amount/use of psychiatric medications for every patient during the first 3 postoperative days.
Postoperative infections (numbers of patients with postoperative infections) | 21 days
  numbers of patients with postoperative infections
Length of stay in hospital | 21 days
  participants will be followed for the duration of hospital stay, an expected average of 3 weeks

OTHER OUTCOMES:
Adverse events related to Solu-medrol | First 3 post OR days
  Number of patients with adverse events
Postoperative pain measured by pain score on the verbal rating scale 0-4 | First 3 post OR days
  Measured by pain score on the verbal rating scale 0-4

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Clemmesen, MD, Principal Investigator — Hvidovre University Hospital
Locations (1):
- Copenhagen University Hospital Hvidovre, department of anesthesiology, Hvidovre, Denmark